CLINICAL TRIAL: NCT04976010
Title: Single Cell Leukocyte Landscapes and Cardiovascular Risk in Children With Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Johannes Benjamin Holle, Dr. med., Charite University, Berlin, Germany
Other Study IDs: EA2/162/17
Record Dates: First submitted 2021-07-03; First posted 2021-07-26 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Chronic Kidney Diseases; Cardiovascular Diseases; Microbial Colonization; Aging
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fecal and blood samples will be collected at a single timepoint at study enrollment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CKD G3-5: Patients with CKD and an estimated eGFR < 60ml/min not yet on dialysis
  Interventions: Other: No intervention
- End stage kidney disease (ESKD) CKD G5 Hemodialysis: Patients on hemodialysis for at least 3 months
  Interventions: Other: No intervention
- Normal kidney function: Patients enrolled with normal kidney function and/or CKD G1 and an estimated eGFR > 90ml/min
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There will be no intervention in the separate goups, as this is an observational study

SUMMARY:
Chronic kidney disease (CKD) is associated with an increased cardiovascular mortality. In particular children with early-onset CKD have a lifelong increased risk to suffer from cardiovascular disease (CVD). Therefore, children with CKD deserve our attention. The immune system in children with CKD is disturbed, exhibiting pro-inflammatory features. Therefore, we aim to learn more about the characteristics of the immune system in early-onset CKD. In this project PBMC of pediatric CKD patients and age-matched healthy controls will be analysed and compared using CITE-Seq as a multimodal scRNAseq phenotyping method. All patients will be clinically characterized to integrate cardiovascular and immunological data.

ELIGIBILITY:
Inclusion Criteria:

* matching to one of the following groups CKD G3-5: estimated eGFR according to Schwartz formula <60ml/min*1,73m2 (no ESKD) CKD G5 D: patients with ESKD treated with hemodialysis for at least 3 months normal kidney function: CKD G1 or no CKD with eGFR > 90ml/min*1,73m2
* informed consent to participate in this study

Exclusion Criteria:

* body weight of less than 15kg
* acute or chronic inflammatory diseases
* fever
* diabetes
* chronic liver disease
* inflammatory bowel disease or other gastrointestinal disorders (constipation, diarrhea, short bowel syndrome)
* antibiotic prophylaxis or treatment within four weeks prior to recruitment

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Only patients treated at the Department of Pediatric Nephrology in Berlin (Charité), Hamburg (UKE) and Leipzig (KfH) will be recruited for this study.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2021-07-17 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
Immunephenotyping of human PBMC | at recruitment
  scRNAseq with Cellular Indexing of Transcriptomes and Epitopes (CITE)-Seq for whole PBMC will be used to gain information on single cell transcriptomes across multiple immune cell populations together with expression levels of classical mmunological surface markers.

SECONDARY OUTCOMES:
Microbiome sequencing of fecal samples | at recruitment
  16S RNA amplicon sequencing and whole genome shotgun sequencing will be perfomred in fecal samples, collected in RNA/DNA shield. This will allow us insights in composition (abundances) and function of the gut microbiome.
Targeted metabolomics of plasma samples | at recruitment
  By using liquid-chromatography (LC) and gas-chromatography (GC) mass-spectrometry plasma samples will be analyzed for tryptophan metabolites and short chain fatty acids (absolute quantifiaction in µM).
Pulse wave velocity | at recruitment
  The pulse wave velocity (m/s) will be measured in all recruited patients by usinfg the Mobilograph. Data will be normalized to age.
Carotid intima media thickness | at recruitment
  The carotid intima media thickness (mm) will be measured using ultrasound imaging of the carotid vessel. Data will be normalized to age.
Echocardiography | at recruitment
  A basic echocardiography will be conducted evaluating diastolic and systolic, right and left ventricular function parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Müller, MD, Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Pediatric Gastroenterology, Nephrology and Metabolic Diseases, Charité-Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No